CLINICAL TRIAL: NCT03456921
Title: Using an End-of-life Conversation Game to Engage Underserved Communities in Advance Care Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: John and Wauna Harman Foundation (Unknown); Hospice Foundation of America (Unknown)
Responsible Party: Principal Investigator, Lauren Van Scoy, Associate Professor of Medicine, Humanities and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Study00009009
Record Dates: First submitted 2018-02-23; First posted 2018-03-07 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Advance Care Planning; Vulnerable Populations; Advance Directives; Terminal Illness
Keywords: health games; community engagement; serious games

STUDY DESIGN:
Intervention Model Description: This project uses an evidence-based and effective intervention--an end-of-life conversation game called "Hello"--to engage and activate participants to perform advance care planning. Quantitative data will be collected before and after immediately playing the game. Focus groups also will be held immediately after the game. Three months to nine months after playing the game, participants will complete surveys and also engage in semi-structured interviews about the game and about their ACP activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Game participants (Experimental): All participants will engage in playing the end-of-life conversation game called "Hello", which involves answering open-ended questions about medical decision making and end-of-life issues.
  Interventions: Other: End-of-life conversation game called "Hello"

INTERVENTIONS:
Other: End-of-life conversation game called "Hello" — To play 'Hello', players are provided 32 open-ended questions in a prearranged order and an equal number of game chips. A player reads aloud the first question. Players then individually write down their answers, and take turns sharing answers with the group (players can opt to pass). Players control how long they share, what they share, and when they are ready to proceed to the next question. During the conversation, players may choose to acknowledge others for a particularly thoughtful, poignant, or even funny comment by giving them a chip. A simple pre-game coin flip determines whether the player with the most chips 'wins' the game ('heads'), or the player with the least amount of chips wins the game ('tails').
  Other Names: Previously named "My Gift of Grace"

SUMMARY:
This national project will provide an effective, evidence-based intervention for advance care planning (ACP) to 50 underserved US communities, those with poor access to healthcare systems due to economic, cultural or other barriers. The project will also examine 15 of the 50 communities to learn about the unique needs of African American communities in regards to ACP and to assess the intervention with this population. The team includes the Hospice Foundation of America and a university-based research team from Penn State Milton S. Hershey Medical Center.

DETAILED DESCRIPTION:
The project goal explores how best to meet the needs of underserved communities to improve engagement in the advance care planning (ACP) process, which is defined as a complex and ongoing process that involves discussions with loved ones and/or clinicians, and/or may involve completion of an advance directive document. This national project involves two components: 1) a community outreach program, Community Game Days; and 2) a research project. The community outreach component seeks to provide an effective, evidence based ACP intervention to 50 underserved communities (defined as those with poor access to healthcare systems due to economic, cultural or linguistic barriers). Of these, 15 African American communities across the United States will be selected for participation in the research aspect of the project which seeks to assess the program's impact on and to learn about the unique needs of African American populations with regard to ACP. A highly integrated, collaborative approach will be used, bringing together a national organization concerned about end-of-life care (the Hospice Foundation of America (HFA) and a university-based academic research team (led by Dr. Lauren Van Scoy at Penn State Milton S. Hershey Medical Center through her research program, Project Talk).

The project teams will organize and support a 14-month long community outreach project that will bring an end-of-life conversation game, "Hello," to 50 communities across the United States. The game has been found to stimulate substantive, enjoyable and meaningful end-of-life discussions among participants. Further, over 70% of participants who played the game went on to perform additional ACP behaviors.2-4 That body of research is limited, however, by a primarily Caucasian or South Asian Indian demographic. It is well established that African Americans have historically low rates of ACP completion when compared to Caucasians and that they often receive overly aggressive and unwanted care at the end-of-life.5,6 Thus, learning how best to engage the African American population in ACP activities is critical. Thus, this research project aims to determine whether and to what extent this priming activity yields similar results in African American communities. The research team will conduct mixed methods research on the impact of the game on the performance of subsequent ACP behavior as well as explore the broad needs of African American communities with regards to ACP.

Fifteen of the 50 qualified locations who can demonstrate through a screening process the ability to attract a majority African American audience will be selected to participate in the research aspect of the project which will involve: 1) pre-game questionnaires to assess population characteristics and readiness to engage in ACP, 2) post- game questionnaires to assess satisfaction, realism about the conversation game and readiness to engage in ACP, 3) post-game focus groups to further explore opinions about the game, the value of priming activities, and the broad needs of the community for encouraging ACP, and 4) 3 month follow-up phone interviews to assess ACP behaviors that have been performed and perceived impact of the priming activity. Participants from the additional 35 sites can opt-in to participate in a 3 months follow-up phone call. As the trial progressed, the time-frame for follow-up phone interviews was extended to 3 - 9 months.

Upon completion of this project, this collaboration is expected to have reached up to 1000 African American individuals and 1,500 other underserved individuals and provided them with an enjoyable and rich experience that facilitates communication about end-of-life issues. The research data is expected to provide a significant contribution to the field by yielding information about the needs of 15 African American communities as well as to yield data related to the impact of the priming activity (the game) on ACP behaviors in this traditionally underserved group.

ELIGIBILITY:
Inclusion Criteria:

1. Are over the age of 18
2. Attend a community Game Day event hosted as part of the Hospice Foundation of America community outreach "Hello Project"

Exclusion Criteria:

1. Do not speak English
2. Have significant difficulties with hearing or speaking difficulties by self-report
3. Do not provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1122 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Rate of ACP Behaviors | 9 months post intervention
  This phone questionnaire assesses whether participants went on to perform various behaviors related to advance care planning.

SECONDARY OUTCOMES:
Change in ACP Engagement Survey scores | Baseline (Day 0); immediately post-intervention (Day 0); 3-9 months post intervention
  This validated questionnaire measure assesses engagement in various ACP behaviors and/or readiness to perform ACP behaviors. Items are scored on a 5 point Likert scale (1-5, with 5 indicating highest readiness to perform ACP). Items are averaged for a final score ranging 1-5.
Conversation satisfaction questionnaire | Immediately post-intervention (Day 0)
  Measures participants' satisfaction with the conversation. There are 5 items in the measure, each item is scored on a 1-7 scale with 1 being lowest conversation satisfaction. The items are averaged for the final score ranging 1-7 with 7 indicating the highest conversation satisfaction.
ACP Values/Beliefs Questionnaire | immediately post-intervention (Day 0)
  Measure participants' attitudes about ACP. This a 8-item questionnaire. Scores are calculated by summative responses and the total score ranges from 7-49 with 7 being the least amount of skepticism (a better outcome).
Conversation Realism Questionnaire | immediately post-intervention (Day 0)
  The Conversation Realism survey is an 8-item questionnaire that measures how realistic players felt the game conversation was. Each question is measured with a 7- point Likert scale, with "1" being the least realistic and "7" being the most realistic (better outcome) conversation.
Net Promoter Score | immediately post-intervention (0)
  The Net Promoter Score is a widely single-question (How likely are you to recommend Hello to friends and family?) used to measure participants' game experience on a 10-point scale. It is measured in two ways: (1) raw score is measured on a 10-point scale with 0 being "not likely at all" to 10 (better outcome) being "extremely likely" (2) calculated score = 10-point scale is broken down as follows: detractor score (0-6); passive score (7-8); promoter score (9-10). Passive scores are ignored. The calculated score is: (total number of promoters) - (total number of detractors) / (total number of responses) = score ranging from - 100 to +100 with +100 being the best (better outcome).
Hello Game Assessment - Qualitative focus group interview | immediately post-intervention (Day 0)
  Group discussions held to collect feedback and opinions about playing the conversation game. Data collected is qualitative.
ACP Needs Assessment - Qualitative focus group interview | immediately post-intervention (Day 0)
  Qualitative focus groups will explore the needs of diverse African American populations with regards to ACP and end-of-life planning

CONTACTS AND LOCATIONS:
Overall Officials: Lauren J Van Scoy, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Hershey College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data may be provided upon request

REFERENCES:
- [Derived] Van Scoy LJ, Green MJ, Witt PD, Bramble C, Richardson C, Putzig I, Toyobo O, Wasserman E, Chinchilli VM, Tucci A, Levi BH. Low Skepticism and Positive Attitudes About Advance Care Planning Among African Americans: a National, Mixed Methods Cohort Study. J Gen Intern Med. 2021 Mar;36(3):705-712. doi: 10.1007/s11606-020-06224-z. Epub 2020 Sep 18. PMID 32948953